CLINICAL TRIAL: NCT06359574
Title: Development and Implementation of a Self-Directed Violence (SDV) Prevention Training Program for the North Carolina Department of Adult Corrections
Brief Title: Core Competency Model for Corrections
Acronym: CCM-C
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: North Carolina Department of Adult Corrections (Unknown); North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Principal Investigator, Robert J. Cramer, PhD, Professor, University of North Carolina, Charlotte
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-24-0209
Record Dates: First submitted 2024-03-06; First posted 2024-04-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Suicide prevention; Self-injury; Risk assessment; Attitudes; Competency; Mental health provider
MeSH Terms: conditions — Behavior; Suicide Prevention; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Competency Model for Corrections (CCM-C) Self-Directed Violence Prevention Training group 1 (Experimental): Receives CCM-C training two weeks after baseline assessment.
  Interventions: Other: Core Competency Model for Corrections (CCM-C) Self-Directed Violence Prevention Training
- Core Competency Model for Corrections (CCM-C) Self-Directed Violence Prevention Training group 2 (Experimental): Receives CCM-C training two weeks after follow-up 1 assessment.
  Interventions: Other: Core Competency Model for Corrections (CCM-C) Self-Directed Violence Prevention Training

INTERVENTIONS:
Other: Core Competency Model for Corrections (CCM-C) Self-Directed Violence Prevention Training — The Core Competency Model (CCM; Cramer et al., 2013, 2019) is an evidence-based educational training program for BHCs in suicide prevention core suicide prevention skills. The ten core competencies are: (1) Manage personal attitudes and reactions to suicide; (2) Maintain a collaborative stance toward the client; (3) Elicit evidence-based risk and protective factors; (4) Focus on current suicide plan and intent of suicidal ideation; (5) Determine risk level; (6) Enact a collaborative evidence-based treatment plan; (7) Notify and involve other persons; (8) Document risk, plan, and reasoning for clinical decisions; (9) Know the law concerning suicide, and; (10) Engage in debriefing and self-care. The CCM will be adapted for this pilot trial. In light of the SDV problem in carceral settings, the CCM for Corrections (CCM-C; Cramer, Kaniuka, & Peiper, 2022) was adapted to address both suicide and self-injury assessment, treatment, and prevention.

SUMMARY:
The overall goal of this project is to design, implement, and revise the Core Competency Model for Corrections (CCM-C), an evidence-based Self-Directed Violence (SDV) prevention training program for correctional mental health providers in the North Carolina Department of Adult Corrections (DAC). The proposed specific aims are:

Aim 1: To create the CCM-C training program. Aim 2: To assess preliminary training effectiveness. Aim 3: To gather training program quality improvement feedback from corrections stakeholders.

DETAILED DESCRIPTION:
Investigators will conduct a pilot feasibility and preliminary effectiveness evaluation of the Core Competency Model for Corrections (CCM-C; Cramer et al., 2022). This training approach involves psycho-educational content, self-assessment tools, interactive exercises to address 10 clinical care and practitioner-focused skill sets for suicide and self-injury risk assessment and management. The protocol employs a waitlist control sequential cross-over design and mixed-method evaluation approach targeting 50-100 NC correctional behavioral health clinicians (BHCs). Through an ongoing academic-community partnership, investigators will employ a Corrections Advisory Panel (CAP) to provide expert review of training. The CAP will comprise six NC-DAC BHCs and 4-6 external BHCs with experience in correctional behavioral health. Two training groups will each provide three assessments via an online self-report evaluation battery gathering information regarding participant demographics; SDV prevention knowledge, attitudes, and perceived skills; incarceration-related attitudes; and perceived importance of and intention to use SDV prevention practices.

ELIGIBILITY:
Inclusion Criteria:

* Behavioral Health Clinician (BHC)
* 18 years of age or older
* Living in the U.S.
* Currently employed by the NC DAC

Exclusion Criteria:

* Decisional or cognitive impairments that preclude being able to consent to study participation
* Being a member of the study correctional advisory panel (CAP)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the CCM-C training intervention | Immediately post-training
  Feasibility of CCM-C training as measured by the Feasibility of Intervention Measure (FIM; Weiner et al., 2017); the scale ranges from 5-20 where higher scores indicate greater feasibility.
Acceptability | Immediately post-training
  Acceptability of CCM-C training as measured by the self-report subscale on the Feasibility of Intervention Measure (FIM; Weiner et al., 2017); the scale ranges from 5-20 where higher scores indicate greater acceptability.
Appropriateness | Immediately post-training
  Appropriateness of CCM-C training as measured by the self-report subscale of the Feasibility of Intervention Measure (FIM; Weiner et al., 2017); the scale ranges from 5-20 where higher scores indicate greater appropriateness.
Usability | Immediately post-training
  Usability of CCM-C training as measured by the self-report subscale of the Feasibility of Intervention Measure (FIM; Weiner et al., 2017); the scale ranges from 5-20 where higher scores indicate greater usability.

SECONDARY OUTCOMES:
Perceived self-directed violence prevention skills | Immediately post-training
  The Suicide Competency Assessment Form (SCAF; Cramer et al., 2013, 2020) will be used to measure participants' perceived SDV prevention skill mastery. The SCAF is a self-report questionnaire that contains 10 items capturing core competencies of the CCM-C training; these items are measured on a four-point scale of perceived competency (1 = incapable; 4 = advanced) where higher scores denote better competency. For the present study, these 10 items was adapted to capture SDV-focused skills.
Willingness to intervene with a suicidal person | Immediately post-training
  The Attitudes about Intervening with a Suicidal Person (AIBS; Aldrich et al., 2014) self-report questionnaire will be used to measure SDV prevention-focused attitudes and the willingness to intervene in an event where a person is experiencing SDV. The AIBS is a subscale of the larger, recently revised Willingness to Intervene against a Suicidal Person Enhanced questionnaire (Aldrich & Cerel, 2023). Higher scores (range 14-90) convey more positive attitudes and greater willingness to intervening with someone in distress.
Beliefs about incarcerated persons engaging in self-directed violence | Immediately post-training
  The Attitudes toward Prisoners who Self-Harm (APSH; Garbutt & Casey, 2015; Ireland & Quinn, 2007) scale is a self-report questionnaire that will be used to measure SDV prevention-focused attitudes and stigma. The APSH consists of 25 items with a total score; higher scores (range 25-125_ denote more stigmatizing beliefs.
Self-directed violence prevention knowledge | Immediately post-training
  For this pilot evaluation, investigators created a 10 multiple-choice CCM-C Knowledge Quiz. Correct answers are summed for a total score (range 0-10) where higher scores indicate greater understanding of the CCM-C.
Perceived importance of training | Immediately post-training
  Investigators will use the intention to use training content scale (Cramer et al., 2019), a brief self-report questionnaire, to capture BHC's perceived importance in using (pre-training) and intent to use (post-training) CCM-C training content. Across seven items, higher scores (item mean 1-5) denote greater perceived importance of the training.

OTHER OUTCOMES:
Compassion fatigue: Job burnout | Immediately post-training
  The Compassion Fatigue-Short Scale (CF-SS; Adams, Boscarino, & Figley, 2006), a self-report questionnaire, will be used to assess feelings of compassion fatigue, conceptualized as secondary traumatic stress (5 items) and job burnout (8 items). This measure contains 13 items. This subscale score denotes higher job burnout (range 8-80).
Compassion fatigue: Traumatic stress | Immediately post-training
  The Compassion Fatigue-Short Scale (CF-SS; Adams, Boscarino, & Figley, 2006), a self-report questionnaire, will be used to assess feelings of compassion fatigue, conceptualized as secondary traumatic stress (5 items) and job burnout (8 items). This measure contains 13 items. This subscale score denotes higher traumatic stress (range 5-50).

CONTACTS AND LOCATIONS:
Locations (1):
- North Carolina Department of Adult Corrections, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cramer RJ, Kaniuka AR, Peiper LJ. The core competency model for corrections: An education program for managing self-directed violence in correctional institutions. Psychol Serv. 2022 Nov;19(4):658-670. doi: 10.1037/ser0000624. Epub 2022 Feb 7. PMID 35130009
- [Derived] Prowten SD, Cacace SC, Moxie J, Peters A, Corral A, Bowman M, Peiper LJ, Cramer RJ. Core competency model self-directed violence prevention training program for corrections: a hybrid feasibility-effectiveness trial. BMC Public Health. 2025 Aug 5;25(1):2655. doi: 10.1186/s12889-025-23853-3. PMID 40764547
- [Derived] Peiper LJ, Cramer RJ, Cacace SC, Peters A, Corral AR, Post AF, Prowten SD, Moxie J. Development and implementation of a self-directed violence prevention training program for correctional behavioral health providers: a clinical trial study protocol. Pilot Feasibility Stud. 2024 Aug 8;10(1):107. doi: 10.1186/s40814-024-01533-0. PMID 39118161

DOCUMENTS (1):
  • Informed Consent Form (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT06359574/ICF_000.pdf